CLINICAL TRIAL: NCT01154933
Title: The Effect of Exenatide on Insulin Requirement, Weight and Inflammation in Obese Type 2 Diabetic Subjects on Insulin
Brief Title: Exeantide in Type 2 Diabetes on Insulin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Principal Investigator, Paresh Dandona, MD, Kaleida Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1930
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- exenatide 5 mcg (Experimental): exenatide 5 mcg
  Interventions: Drug: exenatide 5 mcg
- exenatide 10 mcg (Experimental): exenatide 10 mcg
  Interventions: Drug: exenatide 10 mcg
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: exenatide 5 mcg — exenatide 5 mcg
  Arms: exenatide 5 mcg
Drug: exenatide 10 mcg — exenatide 10 mcg
  Arms: exenatide 10 mcg
Drug: placebo — saline sq
  Arms: placebo

SUMMARY:
Exenatide has been shown to result in better glycemic control in type II diabetes patients. Obesity and diabetes are states of increased inflammation; exenatide is expected to lead to decreased inflammation by virtue of better glycemic control and weight loss.

The purpose of this study is to determine if the addition of Exenatide to diabetic patients will reduce the requirements of insulin particularly the short acting insulin. Exenatide may also lead to decreased inflammation by virtue of better glycemic control and weight loss, or an independent effect.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 20-75 years of age inclusive.
* Type 2 diabetes
* On insulin therapy
* HbA1c ≥7.5% and ≤ 9%
* BMI ≥ 30 kg/m2
* Subjects on statins, ACE inhibitors, metformin, thiazolidinediones and antioxidants will be allowed as long as they are on stable doses of these compounds and the dosage in not changed during the study.

Exclusion Criteria:

* Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous four weeks
* Pregnancy
* Hepatic disease (abnormal LFT's)
* Use of DPP4 inhibitors.
* Renal impairment (serum creatinine > 1.5)
* Participation in any other concurrent clinical trial
* Any other life-threatening, non-cardiac disease
* Uncontrolled hypertension (BP > 160/100 mm of Hg)
* Congestive Heart Failure.
* Use of an investigational agent or therapeutic regimen within 30 days of study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MBBS, Principal Investigator — SUNY at Buffalo
Locations (1):
- Millard Fillmore Gates Hospital, Buffalo, New York, United States

REFERENCES:
- [Derived] Dandona P, Ghanim H, Abuaysheh S, Green K, Dhindsa S, Makdissi A, Batra M, Kuhadiya ND, Chaudhuri A. Exenatide Increases IL-1RA Concentration and Induces Nrf-2-Keap-1-Regulated Antioxidant Enzymes: Relevance to beta-Cell Function. J Clin Endocrinol Metab. 2018 Mar 1;103(3):1180-1187. doi: 10.1210/jc.2017-02343. PMID 29346597

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The exenatide 10mcg group started on 5mcg for a single dose study (samples collected were at 0, 2, 4, and 6 hours)
Groups:
- Exenatide: Period 1 = 5 mcg Period 2 = 10 mcg
Period: Exenatide 5 mcg
Arm/Group | Exenatide | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Exenatide 10 mcg
Arm/Group | Exenatide | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exenatide 10 mcg: exenatide 5mcg and then exenatide 10 mcg
- Total: Total of all reporting groups
Arm/Group | Exenatide 10 mcg | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (3) | 54 (4) | 55 (3)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Data was not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m²] | 39.8 (2) | 39.1 (1.6) | 39.5 (1.8)
HbA1c [Mean (Standard Deviation); unit: %] | 8.6 (0.4) | 8.5 (0.3) | 8.55 (0.4)
Fasting Blood Glucose [Mean (Standard Deviation); unit: mg/dl] | 139 (17) | 128 (13) | 133 (15)
FFA [Mean (Standard Deviation); unit: mM] | 0.69 (0.07) | 0.64 (0.08) | 0.66 (0.08)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Insulin
Description: To compare the fasting insulin level at the end of 12 weeks in patients on exenatide subcutaneously twice daily (5 or 10 mcg/injection) as compared to controls in insulin treated obese type 2 diabetic patients.
Time Frame: after 24 hours fast at baseline and 12 weeks
Measure: Mean (Standard Error); unit: μU/mL
Arm/Group | Exenatide 10 mcg | Placebo
Number analyzed (Participants) | 12 | 12
μU/mL
  At Baseline | 12.7 (2.8) | 13.1 (3.1)
  At 12 weeks | 16.4 (3.2) | 13.9 (5.9)

2. Secondary Outcome: Weight
Description: To compare the body weight at the end of 12 weeks in patients on exenatide subcutaneously twice daily (5 or 10 mcg/injection) as compared to controls in insulin treated obese type 2 diabetic patients
Time Frame: value at 12 weeks minus value at baseline
Measure: Mean (Standard Error); unit: lbs
Arm/Group | Exenatide 10 mcg | Placebo
Number analyzed (Participants) | 12 | 12
lbs | 0 (20) | 3 (18)

3. Secondary Outcome: HbA1c
Description: To compare the HbA1c at the end of 12 weeks in patients on exenatide subcutaneously twice daily (5 or 10 mcg/injection) as compared to controls in insulin treated obese type 2 diabetic patients.
Time Frame: value at 12 weeks minus value at baseline
Measure: Mean (Standard Error); unit: percent
Arm/Group | Exenatide 10 mcg | Placebo
Number analyzed (Participants) | 12 | 12
percent | -1.2 (0.5) | -0.5 (0.3)

4. Secondary Outcome: Intranuclear NFκB Binding Activity
Description: Measured by a gel shift assay showing the NFKB and Oct-1 binding to the doublestranded oligonucleotide containing the NFKB DNA binding site in Exenatide group and placebo group
Time Frame: measured after 6 hours of a single dose of placebo or exenatide treatment for value measured at 12 weeks minus baseline
Measure: Mean (Standard Error); unit: % ratio of NFKB/Oct-1
Arm/Group | Exenatide 10 mcg | Placebo
Number analyzed (Participants) | 12 | 12
% ratio of NFKB/Oct-1 | 26 (7) | 0 (7)

ADVERSE EVENTS:
Description: participants were monitored/assessed for possible adverse events, but none occurred
Groups:
- Exenatide 5mcg Then Exenatide 10 mcg: given exenatide 5mcg followed by exenatide 10mcg
Arm/Group | Exenatide 5mcg Then Exenatide 10 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes